CLINICAL TRIAL: NCT07136025
Title: The Study About the Identification of Treatable Traits of Severe Asthma and the Construction of Personalized Treatment System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Shanxi Bethune Hospital (Other); Henan Provincial People's Hospital (Other); First Affiliated Hospital of China Medical University (Unknown); China-Japan Friendship Hospital (Other); Beijing Tiantan Hospital (Other); Second Xiangya Hospital of Central South University (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KE-347
Record Dates: First submitted 2025-08-18; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-03

CONDITIONS: Asthma
Keywords: treatable traits; asthma; sever; AQLQ; ACQ
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Implement individualized cluster management based on treatable traits
  Interventions: Procedure: Individualized cluster management
- Placebo (Other): Routine asthma treatment according to current guidelines
  Interventions: Procedure: Routine asthma treatment

INTERVENTIONS:
Procedure: Individualized cluster management — Individualized cluster management for treatable traits
  Arms: Intervention group
Procedure: Routine asthma treatment — Routine asthma treatment according to current guidelines
  Arms: Placebo

SUMMARY:
Severe asthma is a complex and heterogeneous disease. Patients with severe asthma can present with different types of airway inflammation, and are often accompanied by a variety of comorbidities and risk factors. Identification of potentially modifiable factors affecting prognosis, that is, "treatable characteristics", and individualized bundle management based on these characteristics may help to improve the quality of life of patients with asthma and improve the level of asthma control. Through joint research, this project aims to evaluate the treatable characteristics of asthma in patients with severe asthma in tertiary hospitals across the country, including lung function, fractional exhaled nitric oxide, blood routine, allergen IgE, chest CT, and a detailed questionnaire. The distribution of treatable characteristics of patients with severe asthma and its impact on the quality of life or asthma control level of patients were investigated. For patients with severe asthma, multidisciplinary consultation and shared decision-making were used to establish an individualized bundle management model based on the treatable characteristics of severe asthma. A 6-month randomized parallel controlled clinical trial was conducted to determine whether this model was superior to conventional management in improving the quality of life or asthma control in patients with severe asthma. The implementation of this project will build a new model of individualized management of severe asthma based on treatable characteristics and improve the management level of severe asthma

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, and <80 years with a definite diagnosis of asthma for at least 6 months
* Patients met the 2024 GINA criteria for severe asthma, which was defined as "uncontrolled" asthma (frequent asthma symptoms, or frequent acute exacerbations) despite high-dose inhaled corticosteroids (ICS) plus long-acting β2-receptor antagonists (LABAs), or worsening of symptoms after slight tapering of high-dose therapy.
* They were willing to accept multi-disciplinary and multi-dimensional evaluation and signed informed consent
* Informed consent was obtained and patients were able to participate in the study and 6-month follow-up according to the protocol

Exclusion Criteria:

* The presence of numerous other lung tissue destructive diseases, such as severe bronchiectasis or pulmonary tuberculosis.
* Chest surgery or abdominal surgery in the past 3 months
* Eye surgery had been performed within the past 3 months
* Myocardial infarction within the previous 3 months
* Anti-tuberculosis treatment is ongoing
* Women who are pregnant and lactating
* Macrolide use within 4 weeks before the screening period
* Treatment with anti-ige, anti-IL-5, or anti-IL-5R within 4 weeks before the screening period
* Inhaled ICS+LABA+ long-acting anticholinergic agent (LAMA) for 4 weeks prior to the screening period 4. Allergy to macrolides
* QTc interval prolongation >480ms
* Taking medications that interact with azithromycin, causing QTc prolongation or existing ECG abnormalities, may lead to arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in asthma quality of life score (AQLQ) at 6 months | 6 months

SECONDARY OUTCOMES:
The change of asthma Control questionnaire (ACQ-5) score | At 6 months
Forced Expiratory Volume in 1 second（FEV1） | At 6 months
  Changes in lung function Forced Expiratory Volume in 1 second（FEV1） from baseline
the number of asthma exacerbations within 6 months | within 6 months

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Beijing Institute of Respiratory Medicine and Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Guangzhou Medical University, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://ginasthma.org/2023-gina-main-report